CLINICAL TRIAL: NCT06881823
Title: NeoPSMA: A Phase I/II, Open-label, Multi-center Study of Neoadjuvant Treatment With [177Lu]Lu-PSMA-R2 (AAA602) and [225Ac]Ac-PSMA-R2 (AAA802) in Adults With Prostate-specific Membrane Antigen (PSMA) Positive High-risk Localized Prostate Cancer (HRLPC) Prior to Radical Prostatectomy and Pelvic Lymph Node Dissection
Brief Title: Study to Assess [177Lu]Lu-PSMA-R2 (AAA602) and [225Ac]Ac-PSMA-R2 (AAA802) in Participants With PSMA-positive HRLPC
Acronym: NeoPSMA
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: The radioligands to be evaluated showed acceptable safety but limited benefit in metastatic prostate cancer
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CAAA802B12101; 2024-516952-17-00 (Other: EU CTIS)
Record Dates: First submitted 2025-02-25; First posted 2025-03-18 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Prostate Cancer
Keywords: High Risk Localized Prostate Cancer; prostate-specific membrane antigen; PSMA; neoadjuvant treatment; adults; radioligand therapies; RLT; AAA602; AAA802; Prostate cancer; Phase 1; Phase 2; high-risk localized prostate cancer; HRLPC; Actinium; Lutetium; gozetotide; Radical Prostatectomy; RP; Pelvic Lymph Node Dissection; PLND
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Lutetium-177; Actinium-225; gallium 68 PSMA-11

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- AAA602 (Active Comparator): AAA602 will be administered as a single intravenous dose. Dose escalation and de-escalation steps will be performed in accordance with the BOIN design.
  Interventions: Drug: AAA602; Drug: Gallium (68Ga) gozetotide; Drug: Piflufolastat (18F); Drug: Flotufolastat F 18; Drug: 18F-PSMA-1007
- AAA802 (Active Comparator): AAA802 will be administered as a single intravenous dose Dose escalation/de-escalation steps will be performed in accordance with the BOIN design.
  Interventions: Drug: AAA802; Drug: Gallium (68Ga) gozetotide; Drug: Piflufolastat (18F); Drug: Flotufolastat F 18; Drug: 18F-PSMA-1007
- Control Arm (No Intervention): No neoadjuvant treatment

INTERVENTIONS:
Drug: AAA602 — [177]Lu-PSMA-R2 Radiopharmaceutical solution for injection/infusion.
  Other Names: Lutetium-177
  Arms: AAA602
Drug: AAA802 — [225]Actinium-PSMA-R2 radiopharmaceutical solution for injection/infusion
  Other Names: Actinium-225
  Arms: AAA802
Drug: Gallium (68Ga) gozetotide — Radioligand Imaging compound. Provided as a kit for radiopharmaceutical preparation of gallium (68Ga) gozetotide. Solution for injection.
  Other Names: Locametz; Illuccix
  Arms: AAA602; AAA802
Drug: Piflufolastat (18F) — Radioligand Imaging compound. Provided as a ready-to-use radiopharmaceutical.
  Other Names: Pylarify; Pylclari
  Arms: AAA602; AAA802
Drug: Flotufolastat F 18 — Radioligand Imaging compound. Provided as a ready to use radiopharamceutical.
  Other Names: Posluma
  Arms: AAA602; AAA802
Drug: 18F-PSMA-1007 — Radioligand Imaging compound. Provided as a ready to use radiopharmaceutical.
  Other Names: Fluorine-18 PSMA 1007
  Arms: AAA602; AAA802

SUMMARY:
The purpose of this trial is to learn more about the effects of AAA602 and AAA802 in men with prostate-specific membrane antigen (PSMA) positive high-risk localized prostate cancer (HRLPC) before surgery to remove the prostate and lymph nodes present in the pelvis area. Lymph nodes are small structures near the prostate that help fight infections. These lymph nodes are removed during surgery because they are a site the disease can spread to.

DETAILED DESCRIPTION:
This Phase I/II study is intended to determine the safety, tolerability, anti-tumor activity, pharmacokinetics, and dosimetry of neoadjuvant treatment with the radioligand therapies (RLT) [177Lu]Lu-PSMA-R2 (AAA602) and [225Ac]Ac-PSMA-R2 (AAA802) before surgery, i.e., radical prostatectomy (RP) and pelvic lymph node dissection (PLND), in participants with Prostate-Specific Membrane Antigen (PSMA)-positive high-risk localized prostate cancer (HRLPC).

Study CAAA802B12101 is a Phase I/II open-label, multi-center study investigating AAA602 and AAA802 as neoadjuvant RLTs before surgery in participants with PSMA-positive HRLPC. In Phase I, participants will be assigned to AAA602 or AAA802 dose escalation cohorts to determine the respective maximum tolerated dose (MTD) and/or the recommended dose for Phase II (RP2D). In Phase II, participants will be randomized to one or two investigational arms, i.e., the RP2D of AAA602 or AAA802, or to the control arm. Therefore, Phase II will have two or three treatment arms. In the control arm, participants will be treated with the standard of care (SoC), i.e., they will not receive any neoadjuvant treatment. Supportive care will be allowed.

Following the last dose of completed RLT, participants will complete a post-treatment imaging/Safety follow-up visit. Upon discontinuation of RLT, participants will complete an end of treatment (EOT) visit prior to the post-treatment imaging/Safety follow-up visit.

If participants undergo surgery, the post-treatment imaging/Safety follow-up visit will be performed before undergoing surgery.

After surgery, participants will complete a post-surgery visit and enter the LTFU. No adjuvant treatment is allowed between surgery and biochemical recurrence (BCR).

The investigational treatments in both Phases I and II are neoadjuvant treatment with AAA602 or AAA802 before surgery (RP and PLND). Surgery is to be performed as per the SoC and is not part of the investigational treatment in this study.

The control treatment in Phase II is SoC, i.e., no neoadjuvant treatment.

ELIGIBILITY:
Inclusion Criteria:

* Adults ≥ 18 years of age.
* Participants must have PSMA-positive disease as assessed by PSMA PET/CT scan using a PSMA imaging agent as protocol instructed, with eligibility being determined by the sponsor's central reading rules.
* Histologically confirmed high-risk adenocarcinoma of an intact prostate, and (a) 1 of the following at diagnosis: Gleason score ≥ 8 and/or PSA ≥ 20 nanogram per milliliters (ng/mL), and/or ≥ cT3a or (b) Gleason score 4+3 and PSA ≥ 20 nanogram per milliliters (ng/mL).
* Adequate organ function:
* Bone marrow reserve:
* White blood cell (WBC) count ≥ 3.0 x 109/L and absolute neutrophil count (ANC) ≥ 1.5 x 109/L.
* Platelets ≥ 75 x 109/L.
* Hemoglobin ≥ 8 g/dL
* Hepatic function:
* Total bilirubin ≤ 1.5 x the institutional upper limit of normal (ULN). For participants with known Gilbert's Syndrome ≤ 3 x ULN is permitted.
* Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 3.0 x ULN
* Albumin > 3.0 g/dL
* Renal function:
* Creatinine clearance ≥ 60 mL/min. Note that participants with findings indicating blockage of urinary outflow are not eligible. No evidence of congenital renal abnormalities with known effect on renal function or voiding abnormalities that may interfere, in the opinion of the principal investigator, with the safe administration of the study treatment.
* An Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) of 0 or 1.
* Indicated to receive radical prostatectomy (RP) and pelvic lymph node dissection (PLND).
* Sexually active participants with female partners of childbearing potential are eligible to participate if they agree to follow one of the following methods of contraception consistently, starting from screening, during the study and for at least 6 months after the last dose of study treatment:
* Are abstinent from penile-vaginal intercourse as their usual and preferred lifestyle (abstinent on a long-term and persistent basis) and agree to remain abstinent.
* Are sterilized (with the appropriate post-vasectomy documentation of the absence of sperm in the ejaculate);
* Agree to use a male condom and have their partner use a highly effective method of contraception (failure rate < 1% per year) as described in Section 8.4.6 when having penile-vaginal intercourse with a woman of childbearing potential who is not currently pregnant, and who agrees to the use of a condom by her partner.
* In addition, participants must refrain from donating sperm starting from Screening, during the study and for at least 6 months after the last dose of the study medication.
* Sexually active participants with a pregnant or breastfeeding partner must agree to remain abstinent from penile-vaginal intercourse; or use a male condom during each episode of penile penetration during the study.

Exclusion Criteria:

* Subjects taking prohibited therapies as described in the protocol
* Any approved or investigational systemic anti-cancer therapy (e.g. chemotherapy, investigational therapy, immunotherapy or biological therapy including monoclonal antibodies) administered for the treatment of HRLPC within 28 days (or 5 times the half-life of that therapy whichever is longer) of the anticipated day C1D1.
* Previous treatment with any approved or investigational radioligand therapy, approved or investigational radioisotopes.
* Prior or concurrent radiation therapy of the prostate, other prostate antineoplastic ablative procedures, or hormonal ablation for prostate cancer.
* Diagnosed with other active malignancies that are expected to alter life expectancy or may interfere with disease assessment. Participants with a prior history of malignancy that has been adequately treated and who have been disease free and treatment free for more than 3 years prior to randomization are eligible, as are participants with adequately treated non-melanoma skin cancer and superficial bladder cancer.

Other protocol-defined Inclusion/exclusion may apply.

Ages: 18 Years to 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2026-06-29 (Estimated); Primary Completion 2030-03-31 (Estimated); Study Completion 2033-06-01 (Estimated)

PRIMARY OUTCOMES:
Number of participants with dose-limiting toxicities (DLTs) (Phase l) | At the end of cycle 1 (each cycle is maximum 6 weeks)
  Incidence and severity of dose-limiting toxicities.
Biochemical recurrence free survival (BFS) (Phase ll) | From the date of surgery until the date of confirmed biochemical recurrence or death due to any cause, whichever occurs first assessed to approximately 60 months
  BFS is defined as the time from the date of surgery until the date of confirmed biochemical recurrence (PSA > 0.2 ng/mL on two readings separated by at least 4 weeks measured at least 8 weeks after surgery).

SECONDARY OUTCOMES:
Biochemical response as measured as Prostate Specific Antigen (PSA)50 (Phase ll) | From screening until the end of neoadjuvant treatment assessed to approximately 6 months
  PSA50 is defined as the percentage of participants who achieved a ≥ 50% decrease (that is confirmed by a second PSA measurement ≥ 4 weeks later) from baseline at the end of neoadjuvant treatment.
Overall Response Rate (ORR) at 12 months after surgery (Phase ll) | at 12 months after surgery
  ORR is the percentage of participants with a response without addition of any new antineoplastic therapy. Antineoplastic therapy is defined as PSA < 0.2 ng/ml as per central lab at month 12 (that is confirmed by a second PSA measurement ≥ 4 weeks later).
Change from baseline in domain scores of the EPIC-26 (Phase ll) | From screening to end of long term follow up assessed up to approximately 66 months
  EPIC-26 (expanded prostate cancer index composite) is a health related quality of life assessment. It contains five symptom domains (urinary incontinence, urinary irritative/obstructive, sexual, bowel, hormonal), scored from 0 (worst) to 100 (best), that can be tracked over time to understand symptom burden and functional outcomes.
Change from baseline on FACT-GP5 item (Phase ll) | From screening to end of long term follow up assessed up to approximately 66 months
  FACT-GP5 (Functional assessment of Cancer Therapy item-GP5) is a health related assessment measuring the overall impact of treatment toxicity. The assessment consists of 1 question - 'I am bothered by side effects of treatment'. The scoring range goes from 0 (not at all) to 4 (very much).
Overall Response Rate (ORR) (Phase l & ll) | Month 12, Month 15, Month 18
  ORR is the percentage of participants with a complete biochemical response without addition of any new antineoplastic therapy other than the study medication (AAA602/AAA802 and/or Radical Prostatectomy (RP) and Pelvic Lymph Node Dissection (PLND)). Antineoplastic therapy is defined as PSA < 0.2 ng/ml as per central lab (that is confirmed by a second PSA measurement ≥ 4 weeks later).
Percentage of participants with a functional response on PSMA PET/CT | From screening until the end of neoadjuvant treatment assessed to approximately 6 months
  Functional response is defined as either complete PSMA response if all PSMA-avid lesions had resolved, a partial response if there was >30% decrease in SUVmax, progressive disease if there was >30% increase in SUVmax, or the presence of new PSMA-avid lesions and stable disease if the response did not meet the criteria for complete, partial, or progressive PSMA-avid disease. The response will be assessed at the end of neoadjuvant treatment with radioligand therapy compared to baseline (Eapen et al 2024).
Percentage of participants achieving pathological complete response (absence of disease) or minimal residual disease (Phase l & ll) | From screening until post-surgery follow up assessed at approximately 7.5 months
  Percentage of participants achieving pathological complete response (absence of disease) or minimal residual disease (Ph I & II) as assessed by local review and independent central review.
Concordance in the evaluation of pathological response between local review and independent central review (Phase l & ll) | From screening until post-surgery follow up assessed at approximately 7.5 months
  Correspondence between local and independent central assessment of participants achieving pathological complete response (absence of disease) or minimal residual disease.
Radiation absorbed doses in organs and tumors of AAA602 (Phase l & ll) | From cycle 1 day 1 until until approximately cycle 2 day 3 (cycle is maximum 6 weeks)
  To evaluate tumor and organs dosimetry of AAA602.
Time concentration profiles and Pharmacokinetics parameters of AAA802 and AAA602 | From cycle 1 day 1 until until approximately cycle 1 day 3 (cycle is maximum 6 weeks)
  Time-concentration profiles and PK parameters of AAA602 and AAA802 (e.g. AUC, Cmax).
Percentage of participants with surgical complications graded according to the Clavien-Dindo classification (Phase l & ll)To evaluate surgical safety (phase l & ll) | From screening until post-surgery follow up assessed at approximately 7.5 months
  Number and severity of complications based on the Clavien-Dindo classification (assessment performed post surgery). The Clavien Dindo Classification is used to rank the severity of a surgical complication. It is based on the type of therapy needed to correct the complication. The scale consists of several grades (Grade I, II, IIIa, IIIb, IVa, IVb and V). Grade I complications being the mildest and V being most significant.
Percentage of participants achieving a complete response to therapy (Phase l & ll) | From screening until end cycle 2 assessed up to 20 weeks (cycle is maximum 6 weeks)
  Percentage of participants achieving undetectable PSA and absence of disease on PSMA PET/CT during neoadjuvant treatment. Complete response to safety is defined as: PSA < 0.1 ng/ml that is confirmed by a second PSA measurement ≥ 4 weeks later; the absence of any PSMA uptake on PSMA PET/CT.
Percentage of participants achieving PSA < 0.2 (Phase l & ll) | From cycle 1 day 1 of post progression treatment to approximately 60 months after surgery
  Percentage of participants achieving undetectable PSA (<0.2) after treatment with AAA802 and AAA602 post biochemical recurrence. PSA < 0.2 is confirmed by a second PSA measurement ≥ 4 weeks later in response to treatment with cycles of AAA602 and/or AAA802 administered following biochemical recurrence after surgery;

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent expert panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data is currently available according to the process described on www.clinicalstudydatarequest.com.
URL: https://www.clinicalstudydatarequest.com